CLINICAL TRIAL: NCT05988320
Title: Comparison of the Effect on Fatigue of the Cancer Patient Caregiver Who Applied Pranayama Breathing Exercise and no Application
Brief Title: The Effect of Pranayama Breathing Exercise on Fatigue in Cancer Patient Caregivers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Data from this study collected
Sponsor: Sanko University (Other)
Responsible Party: Principal Investigator, Zeynep Doğan, Lecturer, Sanko University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SANKOU-HEM-ZD-02
Record Dates: First submitted 2023-08-04; First posted 2023-08-14 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Caregiver; Fatigue
Keywords: CAREGİVER; CANCER; PRANAYAMA; FATİGUE
MeSH Terms: conditions — Fatigue; Neoplasms

STUDY DESIGN:
Intervention Model Description: The caregivers of the patients hospitalized in the medical oncology clinic of the Research Center Mehmet Kemal Dedeman Hematology - Oncology Hospital will be formed. Cancer patient caregivers who meet the inclusion criteria of the study and volunteer to participate in the study will constitute the sample of the study.It is planned to take 30 people per group and 60 people in total.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental: Applications to the Intervention Group (Experimental): Pranayama breathing will be performed by the caregivers of cancer patients in the Medical Oncology clinic for a total of 4 weeks, covering 15-20 minutes every day, for a total of 4 weeks. information will be given about the benefits and benefits, and any questions will be answered. The application steps will be repeated both by explaining and showing, until the caregiver learns, and if there are any points that they cannot do, they will be corrected. When the caregivers are observed to perform the application fully, they will be asked to do the pranayama breathing exercise every day for 4 weeks and will provide the effectiveness and continuity of the application by providing the same researcher 3 days a week (Tuesday, Thursday, Saturday) with a smartphone WhatsApp video call.
  Interventions: Procedure: Pranayama breathing exercise
- Applications to the Control Group (No Intervention): Only the pre-test will be applied to the caregivers of cancer patients in the Medical Oncology clinic in the control group. After the caregiver introduction form and Piper fatigue scale application, no breathing exercises will be performed. Individuals will continue their daily lives. Four weeks later the Piper fatigue scale will be administered again. After the Piper fatigue scale is applied, pranayama breathing exercise training will be given to all control group patients and they will be applied for 2 sessions.

INTERVENTIONS:
Procedure: Pranayama breathing exercise — Pranayama is an important step in yoga, way of life, and is translated as "the science of breathing, breath control, willful breathing". This alternating breathing-out action also balances the sympathetic and parasympathetic nervous systems, giving the person a state of calm, providing relaxation and positively affecting fatigue. Application steps; Right hand Nasika mudra is performed. Nasika mudra is the mudra where the second and third fingers of the right hand are folded into the palm and the other fingers are exposed. Then the right nostril is closed with the first finger of the right hand. Start by breathing through the left nostril. Then the left nostril is closed with the fourth finger and the breath is held. While the left nostril is closed, the right nostril is opened and inhaled. Breathe again through
  Arms: Experimental: Applications to the Intervention Group

SUMMARY:
This research is a randomized controlled experimental study to determine the effect of pranayama breathing exercise applied to caregivers of cancer patients on fatigue.

DETAILED DESCRIPTION:
METHODST: The research will be carried out at Erciyes University Health Practice and Research Center Mehmet Kemal Dedeman Hematology - Oncology Hospital located in Kayseri city center.

Population and Sample of the Research: The population of the research will be the caregivers of the patients hospitalized in the medical oncology clinic of Erciyes University Health Practice and Research Center Mehmet Kemal Dedeman Hematology - Oncology Hospital. Cancer patient caregivers who meet the inclusion criteria of the study and volunteer to participate in the study will constitute the sample of the study.

Sample of the Research: It was calculated by performing power analysis for the sample of the research. In the article titled "Evaluation of fatigue and sleep quality of caregivers of advanced cancer patients", the minimum sample size per group was 22 when the calculation was made as alpha=0.05 and power=0.80, taking into account the pretest-posttest fatigue score averages of the caregivers. It is planned to take 30 people per group Data Collection Form and Tools: The data of the study will be collected through the Caregiver Information Form, Piper Fatigue Scale, Informed Voluntary Consent Form, Eastern Cooperative Oncology Group (for the patient) Performance Scale forms.

Data Collection: Ethics committee, institutional permission and scale usage permission were obtained for the data of the study. Intervention and control group selection in the study will be collected by minimization randomization. The data will be collected by the researcher himself by face-to-face interview method. The intervention group will be given pranayama training. The post-test will be done four weeks after both groups are pre-tested.

Pre-Test: . After informing the caregivers of cancer patients in the Medical Oncology clinic about the research and obtaining verbal and written consent from the researcher, the caregiver introduction form and Piper fatigue scale will be applied to the experimental and control groups, respectively.

Post-Test: The piper fatigue scale will be re-administered to the individuals in both groups by the same researcher four weeks after the pre-test, and one day after the pranayama breathing exercise in the control group and experimental group.

ELIGIBILITY:
Inclusion Criteria:

* 1. Above 18 years old 2. Able to read and write 3. Having sufficient communication skills 4. Does not have any ailment that will reduce the ability to grasp and understand 5. Giving active care to inpatients in the clinic 6. Able to use smart mobile phone 7. Caregivers who agree to participate in the study will be included in the study.

Exclusion Criteria:

- 1. Having a chronic disease 2. Caregivers using opioids or sedating drugs will not be included in the study.

3. Using integrated health practices in the treatment process 4. Patients who exercise regularly will not be included in the study.

Research Termination Criteria

Intervention Group

1. Developing health problems
2. Unwilling to continue Pranayama practice
3. Not practicing pranayama as recommended or unable to do it effectively,
4. The study will be terminated with patients who want to withdraw from the study.

Control Group

1. Developing health problems
2. The study will be terminated with patients who want to withdraw from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2023-03-18 (Actual); Primary Completion 2023-10-20 (Actual); Study Completion 2023-11-10 (Actual)

PRIMARY OUTCOMES:
fatigue of cancer caregivers | four weeks
  Measuring the fatigue of cancer patient caregivers before and after four weeks of training

CONTACTS AND LOCATIONS:
Locations (1):
- Erciyes University, Kayseri, Talas, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
We plan to share it after it is ready for publication.